CLINICAL TRIAL: NCT07294118
Title: Endovascular Infusion of Lidocaine and Steroids in the Middle Meningeal Artery for Pain Management in Spontaneous Subarachnoid Hemorrhage Patients
Brief Title: Infusion of Lidocaine and Steroids in Middle Meningeal Artery for Pain in Subarachnoid Hemorrhage
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-0010
Record Dates: First submitted 2025-05-21; First posted 2025-12-19 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Headache; Opiate Dependence; Opioid Use
MeSH Terms: conditions — Subarachnoid Hemorrhage; Headache; Opioid-Related Disorders | interventions — Lidocaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lidocaine (50 mg bilaterally) (Experimental): The participants will receive 50 mg of lidocaine.
  Interventions: Drug: Lidocaine
- Lidocaine (50 mg) + Dexamethasone (10 mg bilaterally) (Experimental): The participant will receive Lidocaine (50 mg) + Dexamethasone (10 mg bilaterally)
  Interventions: Drug: Lidocaine and Dexamethasone
- No injection (Control group) (No Intervention): The participant will not receive an injection.

INTERVENTIONS:
Drug: Lidocaine — The participants will receive 50 mg of lidocaine.
  Arms: Lidocaine (50 mg bilaterally)
Drug: Lidocaine and Dexamethasone — The participants will receive 50 mg of lidocaine and 10 mg of dexamethasone one after the other.
  Arms: Lidocaine (50 mg) + Dexamethasone (10 mg bilaterally)

SUMMARY:
The goal of this clinical trial is to learn if an infusion of lidocaine, with or without steroids, into the middle meningeal artery (MMA) helps relieve severe headaches in patients with spontaneous subarachnoid hemorrhage (SAH). It will also study the safety of this treatment.

DETAILED DESCRIPTION:
This protocol outlines a single-arm prospective cohort study evaluating the efficacy of endovascular infusion of lidocaine and steroids into the MMA for managing post-SAH pain (i.e., headaches) in patients with SAH with Hunt and Hess Grades 1-2. 15 patients will be enrolled into three groups of treatment: lidocaine, lidocaine/dexamethasone, and no injection. Pain outcomes will be evaluated using VAS at multiple timepoints, including during neurochecks postoperatively, to calculate a cumulative "total VAS score." Morphine equivalents will also be tracked to assess opioid needs over time.

The main questions it aims to answer are:

Does the infusion lower patients' pain levels after SAH?

Does the infusion reduce the amount of opioids and other pain medications patients need?

Are there any side effects or complications from the procedure?

Researchers will compare three groups:

Patients who receive lidocaine alone

Patients who receive lidocaine with dexamethasone (a steroid)

Patients who receive no infusion

All participants will:

Undergo a standard brain angiogram (a routine imaging test for SAH)

May receive the medication during the angiogram, depending on their assigned group

Be monitored closely for changes in pain and medication use

Complete follow-up visits at 1, 3, and 6 months to track outcomes and side effects

This study may help find new, targeted ways to treat headaches in patients with SAH and reduce reliance on opioids.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Diagnosed with aneurysmal SAH, Hunt and Hess Grades 1-2.
* Consent to study procedures and follow-up evaluations.

Exclusion Criteria:

* Known allergies to lidocaine or steroids.
* Arteriovenous malformations.
* Dural Arteriovenous Fistulas.
* Other significant intracranial pathologies.
* Hemodynamic instability preventing safe intervention.
* Previous MMA interventions.
* Previous craniotomies or need for craniotomy.
* Need for external ventricular drain.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Score | Baseline
  The Visual Analog Scale (VAS) is a validated, subjective measure for assessing pain intensity. It consists of a 10-centimeter horizontal line anchored by two extremes: "no pain" (0 mm) and "worst imaginable pain" (100 mm). Participants indicate their pain level by marking a point along the line that corresponds to their current pain intensity. The score is determined by measuring the distance in millimeters from the "no pain" anchor to the participant's mark, yielding a score between 0 and 100 mm. Higher scores represent greater pain intensity.
Visual Analog Scale (VAS) Score | Every 4 hours for 24 hours following the procedure
  The Visual Analog Scale (VAS) is a validated, subjective measure for assessing pain intensity. It consists of a 10-centimeter horizontal line anchored by two extremes: "no pain" (0 mm) and "worst imaginable pain" (100 mm). Participants indicate their pain level by marking a point along the line that corresponds to their current pain intensity. The score is determined by measuring the distance in millimeters from the "no pain" anchor to the participant's mark, yielding a score between 0 and 100 mm. Higher scores represent greater pain intensity.

SECONDARY OUTCOMES:
Analgesic Use by Category and Total Quantity (Non-Opiates) or Morphine Equivalents (Opiates) - Pre- and Post-Intervention | up to 6 months
  To measure analgetic use by category and total quantity in the case of non-opiates, or morphine equivalents in the case of opiates, pre- and post-intervention. by category and total quantity in the case of non-opiates, or morphine equivalents in the case of opiates, pre- and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kan Peter, MD, Principal Investigator — University of Texas Medical Branch, Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Galveston, Texas, United States